CLINICAL TRIAL: NCT06829771
Title: Phase Ib/II Clinical Trial of TQB2825 Injection Combined Immunochemotherapy in Subjects With Diffuse Large B Cell Lymphoma
Brief Title: Clinical Trial of TQB2825 Injection Combined Immunochemotherapy in Subjects With Diffuse Large B Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2825-Ib/II-01
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2825 injection +R-CHOP (Experimental): TQB2825 injection+R-CHOP (Rituximab+Cyclophosphamide+Doxorubicin Hydrochloride+Vincristine+Prednisone) TQB2825 injection,Rituximab,Cyclophosphamide,DoxorubicinHydrochloride,Vincristine,Prednisone,21 days as a treatment cycle.
  Interventions: Drug: TQB2825 injection +R-CHOP regimen
- TQB2825 injection + GemOx (Gemcitabine + Oxaliplatin) (Experimental): TQB2825 injection, Gemcitabine, Oxaliplatin, 21 days as a treatment cycle.
  Interventions: Drug: TQB2825 injection + GemOx

INTERVENTIONS:
Drug: TQB2825 injection +R-CHOP regimen — R-CHOP is a cancer treatment regimen that uses a combination of five drugs to treat non-Hodgkin lymphoma, e.g., Rituximab+Cyclophosphamide+Doxorubicin Hydrochloride+Vincristine+Prednisone (R-CHOP).
  TQB2825 Injection: TQB2825 is a bispecific antibody targeting the cluster of differentiation 20 (CD20) receptor on tumor cells and the cluster of differentiation 3 (CD3) receptor on T cells.
  Rituximab: A monoclonal antibody that binds to the CD20 antigen on the surface of B cells.
  Cyclophosphamide: An alkylating agent that inhibits the synthesis of DNA and proteins in cancer cells.
  Doxorubicin Hydrochloride: An antineoplastic antibiotic that inhibits the synthesis of DNA and RNA.
  Vincristine: A microtubule inhibitor that blocks the normal function of microtubules during cell division.
  Prednisone: A corticosteroid drug with anti-inflammatory, anti-allergic, immunosuppressive, and anti-cancer effects.
  TQB2825 injection + GemOx (Gemcitabine + Oxaliplatin)
  Arms: TQB2825 injection +R-CHOP
Drug: TQB2825 injection + GemOx — TQB2825 Injection: TQB2825 is a bispecific antibody targeting the CD20 receptor on tumor cells and the CD3 receptor on T cells.
  Gemcitabine: A nucleoside analog that inhibits DNA synthesis. Oxaliplatin: A platinum-based chemotherapy drug that forms cross-links with DNA, inhibiting DNA replication and transcription.
  Arms: TQB2825 injection + GemOx (Gemcitabine + Oxaliplatin)

SUMMARY:
To explore the efficacy and safety of TQB2825 injection combined immunochemotherapy in subjects with untreated or R/R DLBCL.

The efficacy evaluation indicators are objective response rate (ORR), complete response rate (CR rate),progression free survival (PFS), duration of response (DOR) and overall survival(OS).

The safety evaluation indicators are dose-limiting toxicity (DLT) , maximum tolerated dose (MTD)and recommended phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study, sign the informed consent form, and have good compliance;
* Age 18 to under 80 years old (calculated from the date of signing the informed consent form);
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2;
* Life expectancy greater than 12 weeks;
* In the dose expansion phase, previously untreated patients with International Prognostic Index (IPI) scores of 2-5;
* A confirmed diagnosis of diffuse large B-cell lymphoma or grade 3b follicular lymphoma, in accordance with the 2022 World Health Organization (WHO) diagnostic criteria, based on histology or cytology (including diffuse large B-cell lymphoma-not otherwise specified and transformed from indolent lymphomas, not allowing for the following types or components: double-hit, triple-hit, or high-grade B-cell lymphoma-not otherwise specified, mediastinal large B-cell lymphoma, T/histiocyte-rich large B-cell lymphoma, human herpesvirus 8 (HHV8)-positive/primary effusion lymphoma, Anaplastic lymphoma kinase (ALK)-positive large B-cell lymphoma, Burkitt's lymphoma, and Hodgkin's lymphoma, etc.);
* Immunophenotypic analysis shows that the tumor is CD20 positive;
* Previous treatment meets the following criteria:

  1. Combined with R-CHOP patients: previously untreated diffuse large B-cell lymphoma patients, allowing for corticosteroid pre-treatment (with or without vincristine) or non-curative palliative local radiotherapy.
  2. Combined with GemOx patients: patients with diffuse large B-cell lymphoma who have received at least one line of systemic treatment (including at least one line with CD20 monoclonal antibody) and are not suitable for hematopoietic stem cell transplantation or have failed treatment after transplantation or relapsed, and whose disease progressed during the most recent treatment or relapsed after completion of treatment or confirmed no objective response after adequate treatment.
* According to the 2014 Lugano criteria, there is at least one measurable lesion, i.e., lymph node lesions with a long diameter >15 mm or extranodal lesions with a long diameter >10 mm based on CT cross-sectional imaging; Positron emission tomography (PET)-computed tomography (CT) scan shows PET positivity;
* Laboratory tests meet the following criteria (not corrected with blood transfusion or hematopoietic growth factors within 14 days before screening):

  1. Hemoglobin (HGB) ≥80g/L;
  2. Absolute neutrophil count (NEUT) ≥1.0×10∧9/L;
  3. Platelet count (PLT) ≥ 75×10∧9/L (if accompanied by bone marrow invasion, platelets ≥50×10∧9/L).
  4. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN. If accompanied by liver metastasis, then ALT and AST ≤ 5 ULN;
  6. Serum creatinine (CR) ≤ 1.5 ULN or estimated glomerular filtration rate ≥50 ml/min by the Cockcroft-Gault formula.
  7. Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR) ≤ 1.5×ULN (not on anticoagulant therapy);
* Women of childbearing age must agree to use effective contraceptive measures during the study and for 12 months after the study ends, with a negative serum or urine pregnancy test within 7 days before study enrollment; men must agree to use effective contraceptive measures during the study and for 12 months after the study ends.

Exclusion Criteria:

* The subject has had or currently has other malignant tumors that occurred within 5 years before the first dose of the study drug. The following two situations are eligible for enrollment: other malignant tumors that have been treated with single surgery and have achieved continuous 5 years of disease-free survival (DFS); cured carcinoma in situ of the cervix, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumors), Tis (carcinoma in situ), and T1 (tumors infiltrating the basement membrane)];
* Adverse reactions from previous treatments have not recovered to a Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade score of ≤1, except for grade 2 alopecia, non-clinically significant and asymptomatic laboratory abnormalities, and hypothyroidism stabilized with hormone replacement therapy, which are deemed to have no safety risks by the investigator;
* Received major surgical treatment, significant traumatic injury within 4 weeks before the first dose, or expected to undergo major surgery during the study treatment period, or has long-term unhealed wounds or fractures;
* Any subject with bleeding or bleeding events ≥CTC AE grade 3 within 4 weeks before the first dose;
* A history of arterial/venous thrombotic events within 6 months before the first dose, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism, or any other history of serious thromboembolism (thrombosis from implanted venous access ports or catheters, or superficial vein thrombosis is not considered "serious" thromboembolism);
* Clinically significant uncontrollable pleural effusion requiring repeated drainage, ascites, moderate or greater pericardial effusion;
* Decompensated cirrhosis (Child-Pugh liver function rating of B or C) and active hepatitis (hepatitis B reference: positive HBsAg, and positive hepatitis B virus (HBV) DNA or detection value exceeding the lower limit of detection; hepatitis C reference: positive HCV antibody, and positive hepatitis C virus (HCV) RNA or detection value exceeding the lower limit of detection); Note: Subjects with hepatitis B who are positive for HBsAg, regardless of whether their HBV DNA is detectable, must continue antiviral treatment (nucleoside analogs recommended) and regularly monitor HBV DNA; for subjects with hepatitis B who are positive for HBcAb but negative for HBsAg, regular monitoring of HBV DNA is required, and prophylactic antiviral treatment is recommended; for hepatitis C subjects, regular monitoring of HCV RNA is required.
* Pulmonary diseases, including any of the following conditions:

  1. Past or present non-infectious pneumonia requiring treatment with corticosteroids (including but not limited to acute respiratory distress syndrome, acute hypersensitivity pneumonia, drug-related pneumonia, bronchospasm, acute interstitial pneumonia, idiopathic pulmonary interstitial fibrosis, etc.);
  2. Past or present chronic obstructive pulmonary disease (COPD), and forced expiratory volume in one second (FEV1) <60% (predicted value);
* Brain or mental abnormalities, including any of the following conditions:

  1. A history of substance abuse that cannot be quit;
  2. Accompanying or past central nervous system disease history, including epileptic seizures, hemorrhagic/ischemic stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, paralysis, aphasia, mental illness, consciousness disturbance, unexplained coma, neuropathy, organic brain syndrome, etc.;
  3. Brain MRI evidence indicating inflammatory lesions and/or vasculitis;
  4. Cerebrovascular accidents, cerebral infarction, etc., within 6 months before the first dose;
* Major cardiovascular diseases, including any of the following conditions:

  1. Heart failure of more than grade II according to the New York Heart Association (NYHA) standards or cardiac ultrasound examination: Left ventricular ejection fraction (LVEF) <50%;
  2. A history of clinically significant ventricular arrhythmias (such as sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes ventricular tachycardia) or arrhythmias requiring continuous antiarrhythmic drug treatment;
  3. A history of myocardial infarction, serious arrhythmias, unstable angina, etc., within 6 months before the first dose;
  4. The Fridericia-corrected QT interval (QTcF) is >450 milliseconds (msec) for males and >470 msec for females (if QTc is abnormal, it can be measured three times continuously with an interval of more than 2 minutes, and the average value can be taken);
  5. A history or family history of congenital long QT syndrome;
  6. Hypertension that cannot be controlled with a combination of two drugs (at least two measurement results are systolic pressure ≥160 mmHg, diastolic pressure ≥100 mmHg);
* Active or uncontrolled infections (≥CTC AE grade 2 infections), including bacterial, fungal, or viral infections (including but not limited to active pneumonia, syphilis, tuberculosis, and Coronavirus disease 2019 (COVID-19), etc. During the screening period, Polymerase chain reaction (PCR) testing or two antigen tests for COVID-19 must be performed (with an interval of at least 24 hours), and the test results must be negative to be eligible. Subjects who do not meet the COVID-19 infection eligibility criteria must fail the screening, and can only be re-screened under the following conditions: asymptomatic subjects at least 10 days after the first positive test result, or symptomatic subjects at least 10 days after the onset of symptoms);
* Renal failure requiring hemodialysis or peritoneal dialysis, history of nephrotic syndrome;
* A history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases;
* Having or having had autoimmune diseases that require treatment, subjects receiving stable replacement therapy for hypothyroidism, and type 1 diabetes can be enrolled.
* Prepared for or having received organ transplantation, or having obvious host-graft reactions, or having received allogeneic hematopoietic stem cell transplantation in the past;
* Need for systemic immunosuppressive treatment, including but not limited to: use of cyclosporine, tacrolimus, etc., within 4 weeks before the first dose, receiving high-dose glucocorticoid therapy (prednisone >30 mg/day or equivalent dose of other glucocorticoids), or receiving any other immunosuppressive treatment. Subjects receiving inhaled or local corticosteroid treatment, or those who have been receiving a stable dose of prednisone <10 mg/day or equivalent dose of other glucocorticoids for systemic treatment for at least 4 weeks before the first dose, or those receiving prophylactic medication to prevent infusion reactions before the administration of the trial medication can be enrolled;
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH);
* For relapsed/refractory patients, previous anti-tumor treatments:

  1. Received chemotherapy, immunotherapy, monoclonal antibody treatment within 4 weeks before the first dose, radiotherapy or small molecule targeted drugs within 2 weeks, or still within the 5 half-lives of the drug (the shortest appearing time shall prevail), the washout period is calculated from the end of the last treatment;
  2. Received traditional Chinese medicine (including Compound Eschar Capsules, Kangai Injection, Kanglaite Capsules/Injection, Aidi Injection, Yanzaizi Oil Injection/Capsules, Xiaocaiping Tablets/Injection, Huachansu Capsules, etc.) with anti-tumor indications approved by the National Medical Products Administration (NMPA) in the drug instructions within 2 weeks before the first dose;
  3. Previously used other antibody drugs targeting both CD3 and CD20;
  4. Received Chimeric antigen receptor T (CAR-T) treatment or other immune cell therapy, or autologous hematopoietic stem cell transplantation (auto-HSCT) within 3 months before the first dose;
  5. Previously received R-GemOx or GemOx treatment;
* Known allergies to excipient components of the study drug.
* Participated in and used other anti-tumor clinical trial drugs within 4 weeks or 5 half-lives before the first dose.
* In the judgment of the investigator, there are situations that seriously endanger the safety of the subject or affect the subject's completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity | Baseline to up to two years
  The occurrence of one or more unacceptable toxicities after administration, which prevents the increase of dosage or the extension of the dosing interval.
Maximum tolerated dose (MTD) | Baseline to up to two years
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to up to two years
  ORR: According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune RECIST (iRECIST), the proportion of subjects whose tumors are evaluated as complete response(CR) and partial response(PR) by subcenter imaging evaluation. It is recorded from the first use of the drug to disease progression or initiation of a new anticancer treatment.
Complete response (CR) | Baseline to up to two years
  The percentage of subjects achieving complete response (CR) according to the Lugano classification criteria of 2014.
Progression-free survival (PFS) | Baseline to up to two years
  The period from the first use of the drug to disease progression or death (whichever occurs first).
Duration of Remission (DOR) | Baseline to up to two years
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first) .
Overall survival (OS) | Baseline to up to five years
  From randomization to the time of death from any cause.
Incidence and severity of adverse events (AEs) | Baseline to up to two years
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug.The nature and severity of adverse events were evaluated according to the National Cancer Institute (NCI) standard for common toxicity criteria (CTC) version 5.0 reactions.
Incidence of serious adverse events (SAEs) | Baseline to up to two years
  It refers to adverse medical events such as death, life-threatening, permanent or serious disability or loss of function, hospitalization or prolonged hospitalization, and congenital abnormalities or birth defects after the subject receives the experimental drug.

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Maanshan People's Hospital, Ma’anshan, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Henan Cancer Hospital Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Canser Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The second Hospital of dalian, Dalian, Liaoning
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan university shanghai cancer center, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shannxi
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - People's Hospital of Tianjin (City), Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality